CLINICAL TRIAL: NCT04593134
Title: The Effect of Home Based Walking Exercise on Fatigue, Anxiety, Depression, Sleep Quality, Circadian Rhythms and Quality of Life in Patients With Gastric Cancer Undergoing Gastrectomy
Brief Title: Effectiveness of Exercise Program in Improving Quality of Life in Patients With Gastric Cancer Undergoing Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-10-006A
Record Dates: First submitted 2020-09-21; First posted 2020-10-19 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Gastric Cancer
Keywords: gastrectomy; fatigue; anxiety; depression; sleep quality; Quality of Life
MeSH Terms: conditions — Stomach Neoplasms; Fatigue; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): A 12-week regimen of home-based walking exercises, comprising walking at a moderate intensity for 40 min, three times a Week.
  Interventions: Behavioral: exercise group
- usual-care group (No Intervention): These participants follows the standard post-surgery follow-up consisting of counseling by dietitians, nurses and doctors.

INTERVENTIONS:
Behavioral: exercise group — exercise education: A 12-week regimen of homebased walking exercises, include moderate intensity for 40 min, three times a week.
  We explained the participants how to perform the exercises, according to an instruction manual for the exercise regimen. Participants were instructed that the exercises would be effective only if they reached 40%-60% of the heart rate reserve, as determined by the Karvonen method, or 13-14 on the RPE.
  Exercise education:
  Weekly telephone or mobile application "LINE" consultations concerning exercise.we discussed whether participants' exercise fulfilled the prescribed intensity, duration, frequency and whether the participants experienced any adverse effects.
  Arms: exercise group

SUMMARY:
This study will investigate the effectiveness of a rehabilitation program in improving fatigue, negative emotions , sleep quality, circadian rhythms and quality of life in patients with gastric cancer undergoing gastrectomy in Taiwan.

Hypothesis:

1. The fatigue in exercise group is significant improving than usual-care group at 1st, 2nd, 3rd, 6th, 12th, 24th and 36th month.
2. The negative emotions in exercise group is significant improving than usual-care group at 1st, 2nd, 3rd, 6th, 12th, 24th and 36th month.
3. The sleep quality in exercise group is significant improving than usual-care group at 1st, 2nd, 3rd, 6th, 12th, 24th and 36th month.
4. The quality of life in exercise group is significant improving than usual-care group at 1st, 2nd,3rd, 6th, 12th, 24th and 36th month.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of a rehabilitation program in improving fatigue, negative emotions , sleep quality, circadian rhythms and quality of life in patients with gastric cancer undergoing gastrectomy in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. After undergoing surgery and clinically diagnosed as gastric cancer.
2. Adults over 20 years old.
3. Hemoglobin (above 10 g/dL).
4. Clear consciousness and could communicate in either Mandarin or Taiwanese, and were not cognitively impaired were included.
5. No lower limb disability and able to walk on their own.

Exclusion Criteria:

1. Suspected or confirmed bone metastasis.
2. Poorly controlled cardiovascular disease such as heart failure, arrhythmia, angina, myocardial infarction, chest pain during activities or rest in the past three months, and valvular heart disease using anticoagulants.
3. Poorly diabetes controlled, glycosylated hemoglobin (HbA1C)>9%, blood sugar higher than 250mg/dl or lower than 80mg/dl.
4. Those with poor blood pressure control, systolic blood pressure greater than 160mmHg or diastolic blood pressure than 100mmHg when quiet, and heart rate is greater than 100bpm when quiet.
5. Diagnosed as recurrent depression.
6. Regular exercise above moderate intensity, such as 150 minutes per week in the past three months.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (EORTC QLQ-C30 ) | baseline (one week after recruited)
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30 ) | 1st month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30) | 2nd month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30) | 3rd month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30) | 6th month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30) | 12th month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30) | 24th month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-C30) | 36th month after recruited
  The EORTC QLQ-C30 :This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-C30 consists of three subscales with 30 questions. The EORTC QLQ-C30 have three subscales in the scale include functioning scales (15 questions), symptom scales (13 questions), and global health status (2 questions). The reliability and validity of Cronbach'α was 0.81-0.94. The functional scale and the global health status , the higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | baseline (one week after recruited)
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 1st month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 2nd month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 3rd month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 6th month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 12th month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 24th month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.
Quality of Life (EORTC QLQ-STO22) | 36th month after recruited
  The EORTC QLQ-STO22:This scale is measured by the respondent self-assessed the frequency of various problems in the past week. The EORTC QLQ-STO22 consists of one subscale with 22 questions.The EORTC QLQ-STO22 scale include symptom scales (22 questions) The Cronbach'α was 0.70-0.94.The lower the score in the symptom scale, the better the quality of life.

SECONDARY OUTCOMES:
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | baseline (one week after recruited)
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total； it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 1st month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total；it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 2nd month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total；it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 3rd month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total； it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 6th month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total； it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 12th month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total； it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 24th month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total； it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
fatigue(Brief Fatigue Inventory-Taiwan , BFI-T) | 36th month after recruited
  The scale is measured by the respondent self-assessed the frequency of various problems with activities of daily living in 24 hours. BFI-T has 9 questions in total； it is a self-reported 11-Point Likert Scale. Retest reliability was 0.89-0.97.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | baseline (one week after recruited)
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 1st month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 2nd month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 3rd month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 6th month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 12th month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 24th month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
Emotional distress( Hospital Anxiety and Depression Scale, HADS) | 36th month after recruited
  Emotional distress including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
sleep quality(Pittsburgh Sleep Quality Index and using Actigraph) | baseline (one week after recruited)
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Actigraph is the gold standard for evaluating sleep disorders. As the name suggests, it is an electrophysiological recording of multiple parameters, including total sleep time(TST), sleep efficiency(SE), and sleep onset latency(SOL) which help to score various sleep stages.
sleep quality(Pittsburgh Sleep Quality Index and using Actigraph) | 3rd month after recruited
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Actigraph is the gold standard for evaluating sleep disorders. As the name suggests, it is an electrophysiological recording of multiple parameters, including total sleep time(TST), sleep efficiency(SE), and sleep onset latency(SOL) which help to score various sleep stages.
sleep quality(Pittsburgh Sleep Quality Index and using Actigraph) | 6th month after recruited
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Actigraph is the gold standard for evaluating sleep disorders. As the name suggests, it is an electrophysiological recording of multiple parameters, including total sleep time(TST), sleep efficiency(SE), and sleep onset latency(SOL) which help to score various sleep stages.
sleep quality(Pittsburgh Sleep Quality Index and using Actigraph) | 12th month after recruited
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Actigraph is the gold standard for evaluating sleep disorders. As the name suggests, it is an electrophysiological recording of multiple parameters, including total sleep time(TST), sleep efficiency(SE), and sleep onset latency(SOL) which help to score various sleep stages.
sleep quality(Pittsburgh Sleep Quality Index and using Actigraph) | 24th month after recruited
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Actigraph is the gold standard for evaluating sleep disorders. As the name suggests, it is an electrophysiological recording of multiple parameters, including total sleep time(TST), sleep efficiency(SE), and sleep onset latency(SOL) which help to score various sleep stages.
sleep quality(Pittsburgh Sleep Quality Index and using Actigraph) | 36th month after recruited
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Actigraph is the gold standard for evaluating sleep disorders. As the name suggests, it is an electrophysiological recording of multiple parameters, including total sleep time(TST), sleep efficiency(SE), and sleep onset latency(SOL) which help to score various sleep stages.
Circadian rhythms(using Actigraph) | baseline (one week after recruited)
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.
Circadian rhythms(using Actigraph) | 3rd month after recruited
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.
Circadian rhythms(using Actigraph) | 6th month after recruited
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.
Circadian rhythms(using Actigraph) | 12th month after recruited
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.
Circadian rhythms(using Actigraph) | 24th month after recruited
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.
Circadian rhythms(using Actigraph) | 36th month after recruited
  Circadian rhythms including 24-h autocorrelation coefficient (r24) and in bed less than out of bed dichotomy index (I<O) collection from actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Study Chair — National Taipei University of Nursing and Health Sciences, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 12 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and receive the authors consent.